CLINICAL TRIAL: NCT06402968
Title: Clevidipine for the Antihypertensive Treatment of Acute Intracerebral Hemorrhage
Acronym: CLUTCH
Status: Recruiting | Type: Observational
Sponsor: Zeenat Qureshi Stroke Institute (Other)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 45002
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhage; Stroke; Hypertension
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hypertension | interventions — clevidipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- designated clevidipine hospitals
  Interventions: Drug: Clevidipine Injection
- designated non-clevidipine hospitals
  Interventions: Drug: Alternate IV Antihypertensive Regimen

INTERVENTIONS:
Drug: Clevidipine Injection — Sites will be trained and instructed to administer IV clevidipine according to Food and Drug Administration label, which recommends starting at 1-2 mg/hour, and then doubling the dose initially at short (90 second) intervals. As the BP approaches the goal, the increase in doses should be less than doubling and the time between dose adjustments should be lengthened to every 5-10 minutes. The desired therapeutic response for most patients occurs at doses of 4-6 mg/hour. Most patients have been treated with maximum doses of 16 mg/hour or less. There is limited short-term experience with doses up to 32 mg/hour, and because of lipid load restrictions, no more than 1000 mL or an average of 21 mg/hour of Clevidipine infusion is recommended per 24-hour period. There is little experience beyond 72 hours at any dose.
  Groups: designated clevidipine hospitals
Drug: Alternate IV Antihypertensive Regimen — The alternate IV antihypertensive regimen would be the institutional standard management at designated "non-clevidipine hospitals". It is expected that most of these sites will be using IV nicardipine, which if administered per FDA label is started at 5 mg/hour and increased by 2.5 mg/hour every 5-15 minutes to a maximum dose of 15mg/hour, until desired BP is reached. Once the goal is reached, then the dose may be reduced to 3 mg/hour.
  Groups: designated non-clevidipine hospitals

SUMMARY:
The aim is to compare the rate of hypertensive subjects with ICH who reach SBP target with stability within 60 minutes of enrollment, among patients treated with IV clevidipine with those treated with alternate IV antihypertensive regimen.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older and less than 90 years.
2. Onset of new neurological deficits within 12 hours at the time of enrollment and IV clevidipine or alternate IV antihypertensive regimen can be initiated within 12 hours of symptom onset.
3. Clinical signs consistent with the diagnosis of stroke, including impairment of language, motor function, cognition, and/or gaze, vision, or neglect.
4. Initial National Institutes of Health Stroke Scale (NIHSS) score of 4 or greater.
5. Total GCS score (aggregate of verbal, eye, and motor response scores) of 5 or greater at enrollment.
6. Computed Tomography (CT) scan of the brain demonstrates intraparenchymal hematoma with manual hematoma volume measurement <60 cc.
7. Admission SBP greater than 150 mmHg but less than 220 mmHg on two repeat measurements at least 5 minutes apart, but no more than 10 minutes apart. The reason for exclusion of ICH patients with initial SBP ≥220 mm Hg is based on a post hoc analysis of ATACH-2, which found that patients with initial SBP ≥220 mm Hg (22.8% of the cohort) reported higher rates of neurological deterioration at 24 hours and renal adverse events until day 7 or discharge in patients treated with intensive SBP reduction compared with standard SBP lowering, without any benefit in reducing hematoma expansion at 24 hours or death or severe disability at 90 days.29
8. Signed and dated informed consent by subject, legally authorized representative, or surrogate before index hospital discharge for data collection and agreement to participate in 90- and 180-day follow up visits.
9. Patients with anticoagulant-related ICH are eligible as long as anticoagulant reversal is concurrently undertaken consistent with AHA/ASA guidelines.
10. Patients who will undergo surgical evacuation consistent with AHA/ASA guidelines or local institutional guidelines are eligible unless surgical evacuation is being performed within 6 hours of initiation of IV clevidipine or alternate IV antihypertensive medication regimen. Ultra-early surgery will necessitate use of anesthetic agents which will confound the effect of IV clevidipine or alternate IV antihypertensive medication regimen. Ultra-early surgery/intervention was not used in the minimally invasive catheter evacuation followed by thrombolysis (MISTIE)/ Clot Lysis: Evaluating Accelerated Resolution of Intraventricular Hemorrhage (CLEAR) trials, which required ICH patients to undergo a repeat CT scan after 6 hours to document absence of any hematoma expansion (with ≤5 mL hematoma growth) compared to a previous CT scan prior to any surgical intervention.34,35
11. Patients requiring external ventricular drainage consistent with AHA/ASA guidelines or local institutional guidelines are eligible.

Exclusion Criteria

1. Time of symptom onset cannot be reliably assessed.
2. Previously known neoplasms, arteriovenous malformation (AVM), or aneurysms.
3. Intracerebral hematoma considered to be related to trauma.
4. ICH located in infratentorial regions such as pons or midbrain (cerebellar ICH is not an exclusion criteria).
5. Subject considered a candidate for immediate surgical intervention by the neurosurgery service.
6. Pregnancy, parturition within previous 30 days, or active lactation.
7. Any history of bleeding diathesis or coagulopathy except anticoagulant related ICH.
8. Platelet count of less than 50,000/mm3.
9. Known sensitivity to nicardipine or clevidipine.
10. Patient's living will precludes aggressive ICU management.
11. Patients with allergies to soybeans, soy products, eggs, or egg products.
12. Defective lipid metabolism such as pathologic hyperlipemia, lipoid nephrosis, or acute pancreatitis if it is accompanied by hyperlipidemia.
13. Patients with severe aortic stenosis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All subjects 18 years or older but less than 90 years old who present to the study sites with clinical symptoms consistent with an ICH demonstrated on brain imaging are to be screened for study eligibility.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Monitoring | 15 minutes
  To compare the rate of hypertensive subjects with ICH who reach SBP target with stability within 60 minutes of enrollment, among patients treated with IV clevidipine with those treated with alternate IV antihypertensive regimen. SBP target with stability is defined as achieving a SBP of less than 150 mm Hg and greater than 130 mm Hg with two subsequent consecutive recordings at least 15 minutes apart that show SBP of less than 150 mm Hg and greater than 130 mm Hg.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Antelope Valley Medical Center, Lancaster, California
  - Cleveland Clinic Martin North Hospital, Stuart, Florida
  - Augusta University-Neuroscience Center, Augusta, Georgia
  - University of Michigan Health-West, Wyoming, Michigan
  - University of Missouri, Columbia, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No